CLINICAL TRIAL: NCT01977339
Title: A Randomized, Double-Blinded, Control Trial to Evaluate the Efficacy of Single Injection Femoral Nerve Block With Liposome Bupivacaine for Postsurgical Analgesia in Subjects Undergoing Unilateral Total Knee Arthroplasty
Brief Title: Efficacy of Single Injection Femoral Nerve Block With Liposomal Bupivacaine for Total Knee Arthroplasty
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: New departmental administration, loss of key study faculty
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-0060
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Total Knee Arthroplasty
Keywords: Femoral Nerve Block; Liposomal Bupivacaine
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liposome Bupivacaine (Experimental): Single injection femoral nerve block of 10 cc of 266 mg liposome bupivacaine with 10 cc of normal saline
  Interventions: Drug: Liposome Bupivacaine
- Bupivacaine (Active Comparator): Single shot femoral nerve block with 20cc of 0.25% bupivacaine
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Liposome Bupivacaine — 10 cc of 266 mg liposome bupivacaine with 10 cc of Normal Saline
  Other Names: Exparel
  Arms: Liposome Bupivacaine
Drug: Bupivacaine — 20 cc of 0.25% bupivacaine
  Arms: Bupivacaine

SUMMARY:
The purpose of this study is to compare the quality and duration of pain relief after a total knee replacement provided by a single shot of standard bupivacaine versus a single shot of liposomal bupivacaine, at the site of the femoral nerve. It is hypothesized that the liposomal bupivacaine formulation will provide more effective pain relief than standard bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥18 years of age
2. Scheduled to undergo primary unilateral TKA under general anesthesia.
3. American Society of Anesthesiology (ASA) Physical Status I-III
4. Able to demonstrate motor function by performing a 20-meter walk, and sensory function by exhibiting sensitivity to cold.
5. Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments.

Exclusion Criteria:

1. Currently pregnant, nursing, or planning to become pregnant during the study or within 1 month after study drug administration.
2. Planned concurrent surgical procedure (e.g., bilateral TKA).
3. Body weight < 50 kg (110 pounds) or a body mass index ≥ 40 kg/m2.
4. Contraindication to any of the pain-control agents planned for postsurgical use (i.e., morphine, hydromorphone, oxycodone, bupivacaine).
5. Previous participation in a liposome bupivacaine study.
6. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
7. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the investigator, could interfere with study assessments or compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Opiate consumption | 72 hours
  Compare the cumulative 72 hour opiate consumption after total knee arthroplasty (TKA)in patients who received a single dose of liposome bupivacaine with those who received a single shot femoral nerve block with 0.25% bupivacaine.

SECONDARY OUTCOMES:
Post-operative VAS scores | 1 hr, 4 hrs, 8 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs
  Patients will be asked to describe the pain intensity under two circumstances: pain at rest, and pain on movement. Postoperative pain intensity will be evaluated using the Visual Analogue Scale (VAS) system at 1, 4, 8, 12, 24, 48 and 72 hours. The VAS used will be the 11 point verbal response pain scale with 0 being no pain at all and 10 being the worst possible pain. The patients will be asked to rate their pain levels using this numeric scale.

OTHER OUTCOMES:
Sensory mapping (temperature) | 72 hours
  Sensation in the distribution of the femoral nerve as assessed by temperature using an alcohol swab (0=no sensation, 1=decreased sensation, 2=normal).
Motor function assessment | 72 hours
  The ability to walk 20 meters unassisted with the optional use of a 4-legged walker at baseline, and at 24, 48 and 72 hours post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Shariat, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St. Luke's-Roosevelt Hospital Center, New York, New York, United States